CLINICAL TRIAL: NCT04603872
Title: Clinical Trial for the Safety and Efficacy of CD19/BCMA-targeted CAR-T Cells Combined With Dasatinib for Patients With Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia, B-cell Non-Hodgkin's Lymphoma and Multiple Myeloma
Brief Title: CAR-T Cells Combined With Dasatinib for Patients With Relapsed and/or Refractory B-cell Hematological Malignancies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DASA001
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory; Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphocytic Leukaemia Refractory; Non-Hodgkin's Lymphoma, Relapsed; Non-Hodgkin's Lymphoma Refractory
Keywords: Acute Lymphoblastic Leukemia; Non-Hodgkin's Lymphoma; Multiple Myeloma; CAR T-cell therapy; Dasatinib
MeSH Terms: conditions — Multiple Myeloma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Recurrence | interventions — Dasatinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Administration of CD19/BCMA Targeted CAR T-cells and dasatinib (Experimental): Dose levels of CAR-T cells are based on clinical trials of similar foreign products. Meanwhile, dasatinib would be combined as the following regimens: 1) Dasatinib preconditioning CAR-T cells during the manufacturing; 2) Dasatinib for the intervention of cytokine release storm after CAR-T cell infusion; 3) Dasatinib for the intervention of neurotoxicities after CAR-T cell infusion; 4) Dasatinib for the phase of CAR-T cell decreasing.
  Interventions: Drug: CD19/BCMA Targeted CAR T-cells and dasatinib
- Administration of CD19/BCMA Targeted CAR T-cells (Experimental): Dose levels of CAR-T cells are based on clinical trials of similar foreign products.
  Interventions: Drug: CD19/BCMA Targeted CAR T-cells

INTERVENTIONS:
Drug: CD19/BCMA Targeted CAR T-cells and dasatinib — Each subject receive CS1 Targeted CAR T-cells by intravenous infusion, and the dasatinib was combined according to the presumed regimens.
  Other Names: Administration of CD19/BCMA Targeted CAR T-cells and dasatinib
  Arms: Administration of CD19/BCMA Targeted CAR T-cells and dasatinib
Drug: CD19/BCMA Targeted CAR T-cells — Each subject receive CS1 Targeted CAR T-cells by intravenous infusion.
  Other Names: CD19/BCMA Targeted CAR T-cells infusion
  Arms: Administration of CD19/BCMA Targeted CAR T-cells

SUMMARY:
A Study of CD19/BCMA-targeted CAR-T Cells Combined With Dasatinib for Patients With Relapsed and/or Refractory B-cell Acute Lymphoblastic Leukemia, B-cell Non-Hodgkin's Lymphoma and Multiple Myeloma.

DETAILED DESCRIPTION:
This is a double-arm, single-center study. This study is indicated for relapsed and/or refractory B-cell acute lymphoblastic leukemia, B-cell non-Hodgkin's lymphoma and multiple myeloma, the selections of dose levels and the number of subjects are based on clinical trials of similar foreign products. 120 patients will be enrolled for this trial. Primary objective is to explore the safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of CD19+ ALL, CD19+ NHL, or BCMA+ MM per the US National Comprehensive Cancer Network (NCCN) Clinical Practice Guidelines (2020.v2);
2. Relapsed or refractory B cell hematological malignancies (meeting one of the following conditions):

   1. CR not achieved after standardized chemotherapy;
   2. CR achieved following the first induction, but CR duration is less than 12 months;
   3. Ineffectively after first or multiple remedial treatments;
   4. 2 or more relapses;
   5. Relapse after hematopoietic stem cell transplantation;
   6. Extramedullary leisions which were ineffective to radiotherapy or chemotherapy;
3. Total bilirubin ≤ 51 umol/L, ALT and AST ≤ 3 times of upper limit ofnormal, creatinine ≤ 176.8 umol/L;
4. Echocardiogram shows left ventricular ejection fraction (LVEF) ≥50%;
5. No active infection in the lungs, blood oxygen saturation in indoorair is ≥ 92%;
6. Estimated survival time ≥ 12 weeks;
7. ECOG performance status 0 to 2;
8. Women of childbearing age had negative pregnancy test during screening period and before administration, and agreed to take effective contraceptive measures at least one year after infusion.
9. Patients volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

Subjects with any of the following exclusion criteria were not eligible for this trial:

1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
3. Pregnant (or lactating) women;
4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
5. Active infection of hepatitis B virus or hepatitis C virus;
6. Concurrent therapy with systemic steroids within 2 weeks prior toscreening, except for the patients recently or currently receiving in haledsteroids;
7. Previously treated with any CAR-T cell product or other genetically-modified T cell therapies;
8. Creatinine >2.5mg/dl, or ALT / AST > 3 times of normal amounts, or bilirubin >2.0 mg/dl;
9. Other uncontrolled diseases that were not suitable for this trial;
10. Patients with HIV infection;
11. Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
B-cell acute lymphocytic leukemia(B-ALL), Overall response rate (ORR) | At Month 1, 3, 6, 12, 18 and 24
  Assessment of ORR (ORR = CR + CRi) at Month 6, 12, 18 and 24
B-ALL, Overall survival (OS) | Up to 2 years after CAR-T cells infusion
  From the first infusion of CAR-T cells to death or the last visit
B-ALL, Event-free survival (EFS) | Up to 2 years after CAR-T cells infusion
  From the first infusion of CAR-T cells to the occurrence of any event, including death, relapse orgene relapse, disease progression (any one occurs first), and the last visit
B cell non-hodgkin's lymphoma (B-NHL), Overall response rate (ORR) | At Week 4, 12, and Month 6, 12, 18, 24
  Assessment of ORR (ORR = CR + PR) per Lugano 2014 criteria
B-NHL, disease control rate (DCR) | At Week 12 and Month 6, 12, 18, 24
  Assessment of DCR (DCR=CR+PR+SD) per Lugano 2014 criteria
Multiple myeloma (MM), Overall response rate (ORR) | At Day 28
  Assessment of ORR at Day 28
MM, Overall survival (OS) | At Month 6, 12, 24
  Assessment of OS at Month 6, 12, 24
Quality of life | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale [For item1-28: max score: 112, min score: 28, higher scores mean a better outcome; for item 28-29: max score: 14, min score: 2, higher scores mean a worse outcome] to measure Quality of life at Baseline, Month 1, 3, 6, 9 and 12
Activities of Daily Living (ADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Activities of Daily Living (ADL) scale (Barthel Index) [max score: 100, min score: 0, higher scores mean a better outcome] at Baseline, Month 1, 3, 6, 9 and 12
Instrumental Activities of Daily Living (IADL) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment of Instrumental Activities of Daily Living (IADL) scale [max score: 56, min score: 14, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12
Hospital Anxiety and Depression Scale (HADS) score | At Baseline, Month 1, 3, 6, 9 and 12
  Assessment using Hospital Anxiety and Depression Scale (HADS) [max score: 42, min score: 0, higher scores mean a worse outcome] at Baseline, Month 1, 3, 6, 9 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang, China